CLINICAL TRIAL: NCT02496754
Title: Follicular Long GnRH Agonist Versus Antagonist Protocol in PCOS Women Undergoing in Vitro Fertilization: a Prospective Randomized Controlled Trial
Brief Title: Follicular Long GnRH Agonist Versus Antagonist Protocol in PCOS Women Undergoing in Vitro Fertilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Yingpu Sun, Director of Reproductive Medical Center, 1st Affilated Hospital, Zhengzhou University, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMCZZU-New protocol
Record Dates: First submitted 2015-07-08; First posted 2015-07-14 (Estimated); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Clinical Pregnancy Rate; Ovulation Induction; IVF
MeSH Terms: interventions — ricin A-GnRH conjugate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- New protocol group (Experimental): Use long term GnRH-a 3.75mg at day 2 of menstrual cycle. Around 30 days later, controlled ovarian hyperstimulation using gonadotropins is initiated.
  Interventions: Drug: GnRH-a
- GnRH-antagonist (Active Comparator): In the GnRH antagonist protocol, Gn was injected from day 2-3 of the menstrual cycle and GnRH antagonist (Cetrotide; 0.25 mg) was added daily from day 6 of stimulation. When 2 dominant follicle ≥ 18 mm or three follicles ≥ 17 mm, recombinant human chorionic gonadotropin (hCG) was injected.
  Interventions: Drug: GnRH-anta

INTERVENTIONS:
Drug: GnRH-a — In experimental group, patients use long term GnRH-a; Patients' serum or follicle fluid will be collected if needed.
  Arms: New protocol group
Drug: GnRH-anta — In control group, patients use GnRH-antagonist. Patients' serum or follicle fluid will be collected if needed.
  Arms: GnRH-antagonist

SUMMARY:
Pituitary down regulation is widely used during in vitro fertilization (IVF) procedures. It can suppress the spontaneous luteinizing hormone (LH) surge, and can also make follicles growth evenly.

At present, standard gonadotropin releasing hormone analogue (GnRH-a) long protocol is used in arou Long term GnRH-a, which is usually used in patients with endometriosis,has been shown to increase IVF outcome by altering endometrial receptivity. Moreover, it is also very convenient because patients do not have to inject GnRH-a daily. In order to make patients feel more comfortable during IVF treatment, the investigators have used a new ovarian stimulation protocol since the beginning of 2015. The investigators give patients long term GnRH-a (3.75mg) once at menstrual cycle D2, and begin the use of Gn to stimulate follicle growth around 30 days later based on the hormone levels and follicle size. In the pilot observational study of several patients, no LH surge occurred during ovarian stimulation.

The aim of this randomized controlled study is to compare the efficiency of this new protocol and standard GnRH-a long protocol in the investigator's center.

DETAILED DESCRIPTION:
The primary outcome is clinical prengancy rate. Secondary outcome is cumulative live birth rate. Other parameters include number of oocytes retrieved, 2 pronucleus (2PN) fertilization rate, high quality embryo formation rate, implantation rate, spontaneous abortion rate, and ectopic pregnancy rate.

ELIGIBILITY:
Inclusion Criteria:

* First IVF cycle;
* With normal ovarian reserve(FSH < 10 mIU/mL; antral follicle count>5);
* With normal uterine.
* PCOS women according to Rotterdam criteria

Exclusion Criteria:

* Pre-implantation genetic diagnosis cycles;
* Oocyte donation or sperm donation cycles.

Ages: 22 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1266 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2024-12 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate | 5 weeks after embryo transfer
  5 weeks after embryo transfer, gestational sac with fetal heart present inside uterus

SECONDARY OUTCOMES:
cumulative live birth rate | 2 years after oocyte retrivial
Number of oocytes retrieved | 1 day at oocyte retrieved day
2 pronucleus (2PN) fertilization rate | 48 hours after oocyte retrieved day
  Number of 2PN/Matured oocytes

CONTACTS AND LOCATIONS:
Overall Officials: Yingpu Sun, M.D, Principal Investigator — Zhengzhou University
Locations (1):
- Reproductive Medical Center, 1st Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sallam HN, Garcia-Velasco JA, Dias S, Arici A. Long-term pituitary down-regulation before in vitro fertilization (IVF) for women with endometriosis. Cochrane Database Syst Rev. 2006 Jan 25;2006(1):CD004635. doi: 10.1002/14651858.CD004635.pub2. PMID 16437491
- [Background] Niu Z, Chen Q, Sun Y, Feng Y. Long-term pituitary downregulation before frozen embryo transfer could improve pregnancy outcomes in women with adenomyosis. Gynecol Endocrinol. 2013 Dec;29(12):1026-30. doi: 10.3109/09513590.2013.824960. Epub 2013 Sep 5. PMID 24006906